CLINICAL TRIAL: NCT05818722
Title: Multicentre Retrospective Analysis of the Characteristics and the Long-term Prognosis of the Bicuspid Aortic Valve
Brief Title: A Multicentre Retrospective Study on Bicuspid Aortic Valve
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other); Nanjing Children's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-671
Record Dates: First submitted 2023-02-21; First posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-02

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid Aortic Valve; Echocardiography; Long-term progress
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Bicuspid Aortic Valve (BAV) is a common congenital heart disease with an incidence ranging from 0.16% in Asians to 2% in Westerners. Asian populations with BAV have different morphological characteristics from those of the Western populations, and further elucidation of these differences will serve as a guide for the treatment and follow-up of Asian patients. Therefore, we conducted this multicentre retrospective study to analysis the clinical features, long-term development and surgical prognosis of BAV .

DETAILED DESCRIPTION:
Bicuspid Aortic Valve (BAV) is a common congenital heart disease with an incidence ranging from 0.16% in Asians to 2% in Westerners, and more than one half of patients require medical or surgical treatment within 20 years of diagnosis. Therefore, early diagnosis and effective treatment can help to reduce the incidence of irreversible cardiac impairment and adverse outcomes such as sudden death. Asian populations with BAV have morphological characteristics that differ from those of the Western populations, and further elucidation of these differences could serve as a guide for the treatment and follow-up of Chinese patients. Based on the above background, We conducted this multicentre retrospective study. We will search for patients diagnosed with BAV by echocardiography or other imaging examinations from December 2021 to October 2022 at Nanjing Gulou Hospital, Jiangsu Provincial Hospital and Nanjing Children's Hospital; collect clinical symptoms, signs and examination results of them; find out the specific surgical plan and time of surgery if they have undergone surgery; follow up for symptoms, medication and reexamin Echocardiography to confirm any endpoint events.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a suspected diagnosis of Bicuspid Aortic Valve by echocardiogram from December 2021 to October 2022

Exclusion Criteria:

* Patients with suspected Bicuspid Aortic Valve not clearly diagnosed by echocardiography and not confirmed by cardiac surgery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Bicuspid Aortic Valve
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
All-cause death | 1 year
  Death from any causes
Cardical mortality | 1 year
  Death due to cardiac disease including MI, arrhythmia, heart failure and aortic lesions

CONTACTS AND LOCATIONS:
Overall Officials: Jing Yao, Phd, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Affiliated Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee M, Sung J, Cho SJ, Choi SH, Cho SW, Oh JK, Park SJ, Kim DK. Aortic dilatation and calcification in asymptomatic patients with bicuspid aortic valve: analysis in a Korean health screening population. Int J Cardiovasc Imaging. 2013 Mar;29(3):553-60. doi: 10.1007/s10554-012-0116-3. Epub 2012 Aug 26. PMID 22923281
- [Background] Movahed MR, Hepner AD, Ahmadi-Kashani M. Echocardiographic prevalence of bicuspid aortic valve in the population. Heart Lung Circ. 2006 Oct;15(5):297-9. doi: 10.1016/j.hlc.2006.06.001. Epub 2006 Aug 17. PMID 16914375
- [Background] Fedak PWM. Bicuspid aortic valve and the specialty clinic: are your patients at risk? Cardiol Young. 2017 Apr;27(3):411-412. doi: 10.1017/S1047951117000282. Epub 2017 Mar 6. No abstract available. PMID 28260551
- [Background] Lo Presti F, Guzzardi DG, Bancone C, Fedak PWM, Della Corte A. The science of BAV aortopathy. Prog Cardiovasc Dis. 2020 Jul-Aug;63(4):465-474. doi: 10.1016/j.pcad.2020.06.009. Epub 2020 Jun 26. PMID 32599028
- [Background] Fernandes JF, Gill H, Nio A, Faraci A, Galli V, Marlevi D, Bissell M, Ha H, Rajani R, Mortier P, Myerson SG, Dyverfeldt P, Ebbers T, Nordsletten DA, Lamata P. Non-invasive cardiovascular magnetic resonance assessment of pressure recovery distance after aortic valve stenosis. J Cardiovasc Magn Reson. 2023 Jan 30;25(1):5. doi: 10.1186/s12968-023-00914-3. PMID 36717885